CLINICAL TRIAL: NCT03279471
Title: Specifying and Treating the Anxiety Phenotype in Autism Spectrum Disorder
Brief Title: Specifying and Treating Anxiety in Autism Research
Acronym: STAAR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1097281
Record Dates: First submitted 2017-08-28; First posted 2017-09-12 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Autism Spectrum Disorder; Anxiety
Keywords: autism spectrum disorder; anxiety; cognitive behavior therapy; functional neuroimaging; STAAR; ASD; MIND Institute; UC Davis; MIND; UCD; autism
MeSH Terms: conditions — Autism Spectrum Disorder; Anxiety Disorders; Autistic Disorder | interventions — Sertraline

STUDY DESIGN:
Intervention Model Description: 3 Arm trial comparing manualized CBT/social skills training versus sertraline versus pill placebo
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: participants do not know what interventions others receive; med arm care providers don't know what interventions their patients receive; assessors don't know what treatments the participants they asses receive
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- CBT/BIACA (Experimental): These participants will receive CBT treatment using Behavioral Interventions for Anxiety in Children with Autism (BIACA). BIACA is an anxiety treatment package designed for children with ASD that includes elements of CBT and social skills training.
  Interventions: Behavioral: CBT/BIACA
- Sertraline (Active Comparator): These participants will receive sertraline
  Interventions: Drug: Sertraline
- Pill Placebo (Placebo Comparator): These individuals will receive a pill placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sertraline — Participants start at 12.5 mg and are increased by 12.5/day every two weeks for 14-16 weeks based on their tolerability to the medication. Dosing is capped at 125mg/day.
  Arms: Sertraline
Behavioral: CBT/BIACA — Participants receive 16 weeks of BIACA therapy.
  Arms: CBT/BIACA
Drug: Placebo — Participants are given a placebo capsule with an administration schedule matching that of the sertraline subjects.
  Arms: Pill Placebo

SUMMARY:
The Specifying and Treating the Anxiety Phenotype in Autism Spectrum Disorder (STAAR) study aims to better characterize the sub-group of children and preadolescents with ASD that exhibit clinically significant anxiety by conducting a 16-week randomized comparative treatment trial of the Behavioral Intervention for Anxiety in Children with Autism (BIACA), the medication sertraline, and placebo in youth with ASD ages 8-14 years old. The study involves 2-3 half day telehealth visits for behavioral and medical assessments, 1-2 lab visits for safety testing, and 1-2 optional fMRI visits. The study provides 16-weeks of anxiety treatment involving weekly BIACA therapy either in-person or through telehealth, or medical check-up visits either at the UC Davis MIND Institute or via telehealth. After study completion a 3 month follow up call is conducted and participants in the placebo group are given the option to participate in an additional study phase with the study treatment of their choice. Study participation can be done remotely through the use of telehealth and local labs, visits to the UC Davis MIND Institute are not required for most participants.

DETAILED DESCRIPTION:
Approximately 40%-80% of children and adolescents with autism spectrum disorder (ASD) exhibit clinically significant anxiety symptoms. These symptoms are associated with increased social deficits, depression, irritability, and stereotyped and self-injurious behaviors. Children and adolescents with anxiety also frequently avoid potentially stressful situations, thereby missing opportunities to learn important new skills. Despite the significant consequences of anxiety symptoms, several critical treatment-relevant issues remain unresolved. First, there is a lack of clarity about how to differentiate ASD and anxiety symptoms. Second, little is known about how anxiety manifests in those with ASD and intellectual disability (ID). Third, the neural substrates of anxiety in ASD are poorly understood. The overarching goal of this project is to investigate these open issues in order to make interventions more precise, more personalized, and more likely to promote positive outcomes -- an objective consistent with the National Institutes of Health (NIH), the Roadmap, Precision Medicine, and Research Domain Criteria Project (RDoC) Initiatives and the Interagency Autism Coordinating Committee (IACC) Strategic Plan, Chapter 4.

While there is no doubt that anxiety is a very serious issue for those with ASD, what to do about this problem is less clear. The search for empirically-validated treatments has begun with multiple small trials providing promising evidence that selective serotonin reuptake inhibitors (SSRIs) and cognitive behavior therapy (CBT) might reduce anxiety in those with ASD. However, this work is in its early stages. There is a great need for large, rigorously designed trials that validate the effectiveness of both medication and CBT, as well as functional neuroimaging studies that identify neural predictors of treatment efficacy and markers of therapy-induced change. Such work holds the potential to help answer the questions posed above and to assist the field in developing more personalized treatments. In Project 1 of the Center for the Development of Phenotype-Based Treatments of Autism Spectrum Disorder, we will conduct a study in children with ASD and clinically significant anxiety ages 8-14 to compare efficacy of these different treatment types.

The overall aims of the study are to better characterize the sub-group of children and preadolescents with ASD that exhibit clinically significant anxiety and fears through a 16-week randomized comparative treatment trial of Behavioral Intervention for Anxiety in Children with Autism (BIACA), sertraline, and placebo in youth with ASD, IQ>50, and clinically significant anxiety as assessed by a PARS score that is greater than or equal to 8. Clinician-administered gold standard assays will be used of traditional DSM (Pediatric Anxiety Rating Scale [PARS] and the Anxiety Disorders Interview Schedule-IV [ADIS-IV]), and nontraditional ASD related anxiety symptoms (Autism Spectrum Addendum to the ADIS [ASDD]), as well as parent reports of potentially overlapping symptoms that complicate the ASD anxiety phenotype. Additionally fMRI will be used to investigate neural predictors of treatment efficacy, markers of treatment induced change, and signatures of anxiety sub-types.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatient boys and girls with ASD between ages 8-14 years at consent.
2. Meets criteria for a diagnosis of ASD.
3. Meets criteria for clinically significant anxiety symptoms as defined by a minimum score of 8 on the PARS Severity Scale.
4. Meets criteria for clinically significant anxiety symptoms as defined by qualifying for diagnosis on 1 or more non-phobia items on the ADIS.
5. The child has a Verbal Comprehension IQ greater than 50 as assessed on the Wechsler Abbreviated Scales of Intelligence or other standardized cognitive measure.
6. Anxiety symptoms are considered the primary mental health problem (i.e., most impairing/distressing)
7. Stable medication regimen for 8 weeks prior to screening visit, including alternative medication, nutritionals, or therapeutic diets.
8. Stable non-psychotherapy regimen for 4 weeks prior to screening visits. Non-psychotherapy regimen may include:

   1. Academic tutoring
   2. Occupational therapy
   3. Speech therapy
   4. School aides
9. Stable psychosocial treatment regimen for 4 weeks prior to screening visits. Allowed psychosocial treatments may include:

   1. School counseling (no more than 60 minutes per week in duration)
   2. Psychotherapy
   3. Social skills training
   4. Applied behavior analysis (ABA) (up to 10 hours per week)

Exclusion criteria:

1. Subject is receiving significant concurrent psychosocial treatment with the primary aim to treat the child's anxiety.

   a. Families will have the option of discontinuing such services to enroll in the study. If a potential participant is receiving non-allowed treatments at the time of the phone evaluation and wishes to discontinue these treatments to enter the study, the patient will be asked to discuss this option with their clinician to determine whether termination would be safe and in the child's best interest. We will not influence the decision patients make with their clinician.
2. History of intolerance to sertraline OR previous unsuccessful treatment with sertraline or other SSRIs judged adequate in dose (per list below) and taken for at least 6 weeks, within the past 12 months.

   1. Sertraline - 100mg/daily
   2. Citalopram or paroxetine - 30mg/daily
   3. Escitalopram - 20mg/daily
   4. Fluoxetine - 20mg/daily
   5. Fluvoxamine - 100mg/daily
3. Current clinically significant suicidal behaviors with intent or plan or individuals who have engaged in suicidal behaviors within 6 months. Study physicians will direct patient to appropriate clinical care if these behaviors are seen.
4. Child has unsuccessful treatment for anxiety using a manualized CBT program within the previous 2 years (at least 10 sessions over a period of less than 1 year conducted by a licensed provider of CBT). This will be determined through parent report, records review and speaking with the clinician if appropriate.
5. Lifetime DSM-5 bipolar disorder, schizophrenia or schizoaffective disorder as assessed by all forms of information (i.e., clinical history, data from the ADIS-IV, etc.).
6. Abnormal laboratory or electrocardiogram results at screening that are in the opinion of the investigator clinically significant and may jeopardize the safety of the study subject.
7. Child has a major neurological disorder or medical illness that requires a prohibited episodic or chronic systemic medication that might interfere with the absorption, distribution, metabolism, or excretion of the study medication places the subject at increased risk, or that would interfere with study participation (e.g., frequent hospitalizations, frequent school absences).
8. Child pregnancy as indicated by history or positive pregnancy test.
9. Inability to safely swallow study medication after pill swallowing education.
10. Child and parent/caregiver who do not speak English.

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 68 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2023-02-22 (Actual); Study Completion 2023-02-22 (Actual)

PRIMARY OUTCOMES:
Change in Pediatric Anxiety Rating Scale | Change from 1 Weeks (pre-treatment) to 17 Weeks (treatment completion), and 29 Weeks (3 month post-treatment follow-up)
  The Pediatric Anxiety Rating Scale (PARS) is a clinician-rated scale assessing anxiety symptoms and the associated severity and impairment in children over the past week. The PARS will be used to assess both immediately pre- and post-treatment anxiety, as well as at a 3 month post-treatment follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Marjorie Solomon, PH.D., Principal Investigator — UC Davis
Locations (1):
- UC Davis MIND Institute, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Leyfer OT, Folstein SE, Bacalman S, Davis NO, Dinh E, Morgan J, Tager-Flusberg H, Lainhart JE. Comorbid psychiatric disorders in children with autism: interview development and rates of disorders. J Autism Dev Disord. 2006 Oct;36(7):849-61. doi: 10.1007/s10803-006-0123-0. PMID 16845581
- [Background] Simonoff E, Pickles A, Charman T, Chandler S, Loucas T, Baird G. Psychiatric disorders in children with autism spectrum disorders: prevalence, comorbidity, and associated factors in a population-derived sample. J Am Acad Child Adolesc Psychiatry. 2008 Aug;47(8):921-9. doi: 10.1097/CHI.0b013e318179964f. PMID 18645422
- [Background] van Steensel FJ, Bogels SM, Perrin S. Anxiety disorders in children and adolescents with autistic spectrum disorders: a meta-analysis. Clin Child Fam Psychol Rev. 2011 Sep;14(3):302-17. doi: 10.1007/s10567-011-0097-0. PMID 21735077
- [Background] White SW, Oswald D, Ollendick T, Scahill L. Anxiety in children and adolescents with autism spectrum disorders. Clin Psychol Rev. 2009 Apr;29(3):216-29. doi: 10.1016/j.cpr.2009.01.003. Epub 2009 Jan 25. PMID 19223098
- [Background] Bishop-Fitzpatrick L, Mazefsky CA, Minshew NJ, Eack SM. The relationship between stress and social functioning in adults with autism spectrum disorder and without intellectual disability. Autism Res. 2015 Apr;8(2):164-73. doi: 10.1002/aur.1433. Epub 2014 Dec 19. PMID 25524571
- [Background] Gillott A, Furniss F, Walter A. Anxiety in high-functioning children with autism. Autism. 2001 Sep;5(3):277-86. doi: 10.1177/1362361301005003005. PMID 11708587
- [Background] Craske MG, Stein MB. Anxiety. Lancet. 2016 Dec 17;388(10063):3048-3059. doi: 10.1016/S0140-6736(16)30381-6. Epub 2016 Jun 24. PMID 27349358
- [Background] Vasa RA, Mazurek MO. An update on anxiety in youth with autism spectrum disorders. Curr Opin Psychiatry. 2015 Mar;28(2):83-90. doi: 10.1097/YCO.0000000000000133. PMID 25602249
- [Background] Sukhodolsky DG, Bloch MH, Panza KE, Reichow B. Cognitive-behavioral therapy for anxiety in children with high-functioning autism: a meta-analysis. Pediatrics. 2013 Nov;132(5):e1341-50. doi: 10.1542/peds.2013-1193. Epub 2013 Oct 28. PMID 24167175
- See also: Learn more or sign up for the study here! — https://studypages.com/s/study-of-anxiety-treatments-in-autism-spectrum-disorder-asd-745682/